CLINICAL TRIAL: NCT05919368
Title: The Shape Regulation Mechanism of Yam Pill on Patients With Sarcopenia Based on Intestine-muscle-brain Axis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fujian University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Zhizhen Liu, associate profession, Fujian University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KFKT-2022-012
Record Dates: First submitted 2023-06-09; First posted 2023-06-26 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Sarcopenia
Keywords: Traditional Chinese medicine; Intestinal flora；cognition
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yam pill (Experimental): It consists of sweet potato, white art and ginseng
  Interventions: Dietary Supplement: Yam pill
- placebo group (Placebo Comparator): It consists of corn starch and dextrin
  Interventions: Dietary Supplement: Yam pill

INTERVENTIONS:
Dietary Supplement: Yam pill — It consists of sweet potato, white art and ginseng

SUMMARY:
The main manifestation of sarcopenia is the decline of muscle strength, quality, and physical function, and it has the characteristics of overlapping, changing, or transforming with cognitive and emotional problems， belonging to the category of physical and mental diseases. At present, the effective treatment and mechanism of the disease are still unclear. The team's preliminary study found that the Jingfang Yam pill has unique advantages in "spleen dominates muscle", which can significantly improve the skeletal muscle mass, strength, and endurance of mice. The intestine-muscle-brain axis-spleen deficiency may be the key pathogenesis of sarcopenia. As such, the study proposes a hypothesis: whether Yam pills intervene in patients with sarcopenia is achieved bidirectional balance regulation of the body through the bidirectional communication pathway of the muscle-brain axis regulated by the intestinal flora. This project applies a randomized, placebo-controlled, double-blind RCT study design, with sarcopenia patients as the research objects, and utilizes musculoskeletal ultrasound, gut microbiota, untargeted metabolomics, functional near-infrared imaging, and other multidisciplinary techniques. To explore the mechanism of Yam pill regulating patients with sarcopenia by regulating intestinal microecology and metabolism-related molecules mediated by the "intestine-muscle-brain axis".

DETAILED DESCRIPTION:
This randomized, double-blind, placebo-controlled study intends to recruit 136 qualified sarcopenias with spleen-asthenia syndrome. The trial will be conducted at the Second People's Hospital Affiliated to Fujian University of Traditional Chinese Medicine in Fujian Province, China. All subjects will be required to fill in baseline information before enrollment to determine the general situation of patients before randomization. Subsequently, the subjects were randomly divided into two groups in a 1:1 ratio: the yam pill group (n = 68) and the placebo group (n =68), randomized sequences were provided by statistical experts who were not involved throughout the trial. Among them, the yam pill is a traditional Chinese medicine formula pill composed of yam, white art, and ginseng, and the placebo is mainly composed of corn starch, which is entirely consistent with the appearance, shape, size, color, specification, packaging and label of yam pill. The Chinese medicine formulations of the two groups were provided in the form of a pill and rice soup delivery (3 times a day, 5 days/week, a total of 24 weeks). In addition, to improve patient compliance during the intervention period, patients in both groups were required to attend a health education lecture once a month, and both groups were followed up for 24 weeks after the intervention.

The four-time points were compared before the intervention (0 weeks), during the intervention (after the end of the 12th week), at the end of the intervention (after the end of the 24th week), and during the follow-up (after the end of the 48th week). The main index was the changes in muscle mass ( 24 weeks minus baseline), and the secondary index was the changes in muscle strength (grip strength; 5 times chair stand test); Physical function (e.g. 6-min walking test, gait speed, time-up-go-test); cognitive function, quality of life and clinical efficacy of traditional Chinese medicine were investigated with the forms of questionnaires to explore the clinical effectiveness of yam pills on patients with spleen asthenia syndrome. Secondly, near-infrared spectral imaging (fNIRS) was used to explore whether the improvement of clinical efficacy caused by yam pills after 24 weeks of intervention was related to the hemodynamic changes in the prefrontal cortex and motor cortex brain region based on the dual task of motor cognition. Subsequently, 16S-rRNA sequencing and non-targeted metabolomics were used to explore whether the improvement of clinical efficacy caused by Yam pills after 24 weeks of intervention was related to the regulation of intestinal flora and its metabolites, to finally clarify the musculus-brain crosstalk during the intervention process and explore its potential mechanism of action.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥60 years old, in line with the AWGS diagnostic criteria for sarcopenia, and in line with the TCM dialectical standard of spleen deficiency syndrome;
2. Be able to understand and cooperate with the test, and voluntarily sign the informed consent.

Exclusion Criteria:

1. Motor dysfunction caused by severe nervous system diseases, musculoskeletal system diseases osteoporosis, severe osteoarthritis;
2. severe heart, lung or mental illness, uncontrolled endocrine or metabolic disease, or severe liver or kidney function (such as cirrhosis, a history of kidney stones, kidney failure or dialysis);
3. Inability to communicate properly with the researcher due to speech or uncorrected hearing impairment;
4. Severe cognitive impairment (brief mental state examination: MMSE score < 24 points), unable to understand the content included in the questionnaire and scale;
5. Use of growth hormone, estrogen, progesterone or testosterone supplements for nearly 3 months, or severe nutritional deficiencies;
6. Participate in other trials or Chinese medicine supplement trials in the past three months.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2023-09-12 (Estimated); Primary Completion 2023-09-15 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline muscle mass at 6 months | baseline，After 12 weeks of intervention, after 24 weeks of intervention, and after 24 weeks of follow-up
  Double X-ray absorptiometry (DXA) was used to determine the skeletal mass (AMS) of the limbs of the patients. This method can accurately measure the total and local skeletal muscle mass, adipose tissue mass and bone mass, and calculate the muscle index = AMS/height 2 (kg/m2).

SECONDARY OUTCOMES:
Change from Baseline handgrip strength at 6 moths | After 12 weeks of intervention, after 24 weeks of intervention, and after 24 weeks of follow-up
  Grip strength was assessed using upper limb muscle strength. Using a spring-type grip device, subjects were asked to extend their elbows in a standing position and perform the maximum force isometric contraction with the dominant hand or both hands respectively, repeated three times, with each interval of 1min rest, and the maximum reading was selected as the final grip strength value
Change from Baseline physical performance at 6 moths | After 12 weeks of intervention, after 24 weeks of intervention, and after 24 weeks of follow-up
  The following indicators of physical performance will be evaluated：gait speed(meter/second), 6-minute walking test (meter), short physical performance battery (score),Time Up Go testing (seconds).Among them, the faster the walking speed, the better, the longer the walking distance, the better, the shorter the walking time
Change from Baseline cognition at 6 moths | After 12 weeks of intervention, after 24 weeks of intervention, and after 24 weeks of follow-up
  Scales: Montreal Cognitive Assessment (score), Stroop color words test, and Test of attentional performance，the higher the scale score, the better.
Change from Baseline 16s rRNA at 6 moths | After 12 weeks of intervention, after 24 weeks of intervention, and after 24 weeks of follow-up
  16S rRNA amplification sequencing was used to detect intestinal microbiota, and fecal samples were collected before baseline randomization, after the end of the intervention at week 12 (mid-term assessment), and after the end of the intervention at week 24. Fecal samples will be collected within 1h, and the collected fecal samples will be sorted into 1.8ml sterile frozen tubes with marks on the ice, and the liquid nitrogen will be immediately frozen in the -80℃ refrigerator.
Change from Baseline hemodynamics at 6 moths | After 12 weeks of intervention, after 24 weeks of intervention, and after 24 weeks of follow-up
  The hemodynamic changes of the prefrontal cortex and bilateral motor cortex were measured by functional near-infrared spectroscopy
Change from Baseline small molecule metabolomics at 6 moths | After 12 weeks of intervention, after 24 weeks of intervention, and after 24 weeks of follow-up
  About 5ml of venous blood samples were collected from the subjects in the fasting state in the morning (fasting for 8-10 hours), injected into a test tube containing anticoagulant, mixed, left at room temperature for 30 min, centrifuged at 3000 r/min for 10 min, and the upper serum was taken, numbered and stored in a refrigerator at -80℃ to be measured. It was detected by an automated biochemical analyzer (Mindary, BS-820, Shenzhen, China), and a non-targeted metabolomics method based on ultra-high performance liquid chromatograph-Quadrupole time-of-flight mass spectrometry (UPLC-QTOF-MS) was used to search for differential metabolites before and after sarcosis intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Zhizhen ZZ Liu, Principal Investigator — Fujian University of Traditional Chinese Medicine
Locations (1):
- Suzhou Panomix biomedical tech Co., LTD, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No